CLINICAL TRIAL: NCT00000233
Title: Alternate Day Buprenorphine Administration, Phase X
Brief Title: Alternate Day Buprenorphine Administration, Phase X - 15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-15; R01-06969-15
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1995-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine how subjects will make changes in the amount of medication received when given a monetary alternative to buprenorphine.

ELIGIBILITY:
Please contact site for information.

Ages: 34 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1993-05

PRIMARY OUTCOMES:
Opioid withdrawal
Subjective dose estimate
Drug effect characteristics: ARCI
Money choice

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Petry, Bickel (in press) Buprenorphine self-administration in buprenorphine-maintained, opioid-dependent outpatients: Effects of an alternate reinforcer. Psychopharmacology. Petry, Bickel (in press) Buprenorphine self-administration in buprenorphine-maintained, opioid-dependent outpatients: Effects of an alternate reinforcer. Psychopharmacology
- [Derived] Antoniotti C, Germani MM, Rossini D, Lonardi S, Pietrantonio F, Santini D, Marmorino F, Allegrini G, Daniel F, Raimondi A, Borelli B, Zaniboni A, Conca V, Abraham J, Spetzler D, Maiello E, Boccaccino A, Passardi A, Giordano M, Tamburini E, Korn MW, Masi G, Cremolini C. FOLFOXIRI and bevacizumab in patients with early-onset metastatic colorectal cancer. A pooled analysis of TRIBE and TRIBE2 studies. Eur J Cancer. 2022 May;167:23-31. doi: 10.1016/j.ejca.2022.02.031. Epub 2022 Mar 30. PMID 35366570